CLINICAL TRIAL: NCT01353404
Title: Relative Bioavailability Study of Lipidil® Supra (Fenofibrate 160mg) Versus SYO-0805 (Fenofibrate 65mg) in Normal Healthy Subjects
Brief Title: Relative Bioavailability Study of Lipidil® Supra (Fenofibrate 160mg) Versus SYO-0805 (Fenofibrate 65mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYO0805
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- fenofibrate 65mg, fed condition, per oral (Experimental)
  Interventions: Drug: Sequence 1; Drug: Sequence 2; Drug: Seqeunce 3; Drug: Sequence 4; Drug: Sequence 5; Drug: Sequence 6
- fenofibrate 65mg, fasting condition, per oral (Experimental)
  Interventions: Drug: Sequence 1; Drug: Sequence 2; Drug: Seqeunce 3; Drug: Sequence 4; Drug: Sequence 5; Drug: Sequence 6
- fenofibrate 160mg, fed condition, per oral (Active Comparator)
  Interventions: Drug: Sequence 1; Drug: Sequence 2; Drug: Seqeunce 3; Drug: Sequence 4; Drug: Sequence 5; Drug: Sequence 6

INTERVENTIONS:
Drug: Sequence 1 — fenofibrate 65mg, fed condition, per oral → fenofibrate 65mg, fasting condition, per oral → fenofibrate 160mg, fed condition, per oral
Drug: Sequence 2 — fenofibrate 65mg, fed condition, per oral → fenofibrate 160mg, fed condition, per oral → fenofibrate 65mg, fasting condition, per oral
Drug: Seqeunce 3 — fenofibrate 65mg, fasting condition, per oral → fenofibrate 160mg, fed condition, per oral → fenofibrate 65mg, fed condition, per oral
Drug: Sequence 4 — fenofibrate 65mg, fasting condition, per oral → fenofibrate 65mg, fed condition, per oral → fenofibrate 160mg, fed condition, per oral
Drug: Sequence 5 — fenofibrate 160mg, fed condition, per oral → fenofibrate 65mg, fed condition, per oral → fenofibrate 65mg, fasting condition, per oral
Drug: Sequence 6 — fenofibrate 160mg, fed condition, per oral → fenofibrate 65mg, fasting condition, per oral → fenofibrate 65mg, fed condition, per oral

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of Lipidil® Supra (fenofibrate 160mg) versus SYO-0805 (fenofibrate 65mg) in single dose oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 20-50 years of age
* Weight more than 55kg and within ±20% IBW(Ideal Body Weight)
* Voluntary written informed consent

Exclusion Criteria:

* History or presence of significant renal, neurologic, pulmonary, endocrine, hematology, oncology, urologic, cardiovascular, musculoskeletal or psychiatric disease
* Drug allergies to fenofibrate
* Recent history or evidence of drug abuse
* Recent participation(within 2months) in other clinical studies
* Recent donation of blood(within 2months) or plasma(within 1months)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of Lipidil® Supra (fenofibrate 160mg) versus SYO-0805 (fenofibrate 65mg) | 23 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., M.B.A., Principal Investigator — Clinical Research Institute, Seoul National University Hospital
Locations (1):
- Clinical Research Institute, Seoul National University Hospital, Seoul, South Korea